CLINICAL TRIAL: NCT05245513
Title: Developing and Testing an Intervention to Enhance Recovery Capital Amid Opioid Use Disorder Pharmacotherapy: A Pilot Randomized Trial of Linkage to Recovery Support Services
Brief Title: Enhancing Recovery Capital Amid Opioid Use Disorder Pharmacotherapy: A Pilot Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lauren Hoffman, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P003720
Record Dates: First submitted 2022-02-04; First posted 2022-02-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Community Center Linkage (RCCL) (Experimental): The RCCL arm will involve a brief (~20 minutes) meeting with a recovery coach (i.e. linkage manager), in which the recovery coach will inform the participant of recovery support services, including recovery community centers, and link them to a recovery community center, with the aid of a facilitated connection to a volunteer recovery community center member (i.e. peer facilitator). The linkage manager will also provide the participant with a list of recovery support service resources.
  Interventions: Behavioral: Recovery Community Center Linkage (RCCL)
- Control Condition (CC) (Active Comparator): The CC arm will involve a time-matched meeting with a recovery coach (i.e. linkage manager), in which the recovery coach will broadly inform the participant of recovery support services, including recovery community centers, and provide them with a list of recovery support service resources.
  Interventions: Behavioral: Control Condition (CC)

INTERVENTIONS:
Behavioral: Recovery Community Center Linkage (RCCL) — A certified recovery coach will meet with participants to educate them on recovery support services, including recovery community centers, and link them to a recovery community center, with the aid of a facilitated connection to a volunteer recovery community center member (e.g., calling a standby peer, scheduling a meet-up at the center). The coach will also provide the participant with a brochure of recovery support resources.
  Arms: Recovery Community Center Linkage (RCCL)
Behavioral: Control Condition (CC) — A certified recovery coach will meet with participants to educate them on recovery support services more broadly, including recovery community centers, and will provide them with a brochure of recovery support resources.
  Arms: Control Condition (CC)

SUMMARY:
The aims of the current study are to: Aim 1. Develop and refine a novel intervention protocol for individuals receiving medication treatment for opioid use disorder that assertively links them to recovery community centers; Aim 2. Determine the feasibility, acceptability, and preliminary efficacy of assertive linkage to recovery community centers relative to a matched control condition, via a pilot randomized controlled trial; Aim 3. Explain quantitative findings by gaining an in-depth understanding of the intervention's feasibility, acceptability, and preliminary efficacy via qualitative interviews.

DETAILED DESCRIPTION:
This 5-year project seek to advance our understanding of the clinical and public health utility of recovery community centers and help bridge the gap between clinical treatment and community-based recovery support services. As a first step in this work, the investigators will develop and test a new intervention for peer-facilitated assertive linkage of patients receiving opioid use disorder pharmacotherapy to recovery community centers (RCCL), relative to a matched control condition (CC). This study aims to: Aim 1. Develop, manualize, and refine RCCL and CC protocols via stakeholder feedback. RCCL and CC protocols will be developed and manualized by adapting published community-based mutual-help linkage protocols. Upon preliminary manual development, feedback cycles will be conducted with relevant stakeholders (recovery coaches, recovery community center members, pharmacotherapy prescribers) to inform protocol revision, and promote its feasibility, acceptability, and adoptability. Aim 2. Determine the feasibility, acceptability, and preliminary efficacy of RCCL versus CC, via a pilot randomized controlled trial. More specifically, the feasibility of study procedures and RCCL/CC interventions, acceptability of interventions, and preliminary efficacy of RCCL relative to CC will be assessed. Aim 3. Explain quantitative findings by gaining an in-depth understanding of RCCL feasibility, acceptability, and efficacy via qualitative interviews in a subset of RCCL participants, peer facilitators, and linkage managers.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* past-year opioid use disorder diagnosis per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
* currently undergoing outpatient buprenorphine treatment through a provider or program at Massachusetts General Hospital
* current residence in Massachusetts

Exclusion Criteria:

* non-English fluency
* active suicidality
* neurodevelopmental disorders or neural trauma preventing informed consent
* active psychosis
* past-year attendance at a recovery community center or recovery support center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall recruitment feasibility | Through study completion, ~3 years from recruitment initiation
  Number of participants successfully recruited within allotted recruitment time frame (~3 years)
Overall intervention feasibility | From the date of intervention manual finalization until the date of study completion, assessed up to 48 months
  Assessed via the Feasibility: Intervention Implementation & Training scale average total score. This is a 2-item instrument to assess perceived intervention feasibility. Items are measured on a 6-point Likert scale (Strongly Disagree-Strongly Agree). Score is the calculated mean. Higher scores indicate greater feasibility.
Fidelity: Linkage manager adherence | From date of first linkage manager meeting until the date of last linkage manager meeting, assessed up to 36 months
  Percent adherence of linkage managers to intervention protocols, as evaluated by the percentage of sessions that are scored with adequate adherence and assessed by recordings of intervention delivery and adherence evaluation materials developed as part of Aim 1 (e.g., adherence rating scales of critical topics). This is a 14-item instrument evaluating the extensiveness of linkage managers' delivery of critical intervention topics. Items are measured on a 5-point Likert scale (Not at all - Extensively). Score is the calculated mean. Total scores range from 1 to 5, with scores > 3 indicating adequate adherence.
Overall intervention acceptability | Month 1
  Assessed via 1 single-item statement addressing the the acceptability of the intervention. The item is measured on a 6-point Likert scale (Strongly Disagree - Strongly Agree). Higher scores indicate greater acceptability.
Overall intervention satisfaction | Month 1
  Assessed via the Client Satisfaction Questionnaire-8 (CSQ8) total score. This is an 8 item measure of client satisfaction with services. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.
Recovery community center attendance | From the date of linkage manager meeting until the date of month-3 follow up, assessed up to 3 months
  Percent of participants who attended a recovery community center 1+ time post linkage manager meeting, as assessed via the Timeline Follow Back
Use of recovery support services | From the date of linkage manager meeting until the date of month-3 follow up, assessed up to 3 months
  Percent days use of any recovery support services post linkage manager meeting, as assessed via the Timeline Follow Back

SECONDARY OUTCOMES:
Participant retention | From the date of first participant enrollment in the trial to the date of study completion, up to 42 months
  Percent of enrolled participants who complete Month 3 Follow-Up
Feasibility of peer facilitator meet-ups | Month 1; Month 3
  Percent of peer facilitator meet-ups occurring within 2 weeks of participant's linkage manager meeting
Intervention appropriateness | Month 1
  Assessed via the Intervention Appropriateness Measure (IAM; adapted for study parameters) average total score. This is a 4-item instrument to assess perceived intervention appropriateness. Items are measured on a 5-point Likert scale (Strongly Disagree-Strongly Agree). Score is the calculated mean. Higher scores indicate greater appropriateness.
Intervention helpfulness | Month 1; Month 3
  Assessed via 4 single-item statements addressing the intervention's helpfulness in general and helpfulness to supporting treatment and opioid use disorder recovery. Items are measured on a 6-point Likert scale (Strongly Disagree-Strongly Agree). Score is the response for each item. Higher scores indicate greater helpfulness.
Change in recovery capital from baseline to Month 3 | Baseline; Month 1; Month 3
  Assessed via the REC-CAP Inventory total score. Scores range from -100 to +100, with higher scores indicating greater recovery capital.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No